CLINICAL TRIAL: NCT05915832
Title: Effects of Remote Ischemic Conditioning on Cerebral Hemodynamics in Patients With Ischemic Stroke(RICCH-IS)
Brief Title: Effects of Remote Ischemic Conditioning on Cerebral Hemodynamics in Patients With Ischemic Stroke
Acronym: RICCH-IS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Vice President of The First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RICCH-IS
Record Dates: First submitted 2023-06-06; First posted 2023-06-23 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC (Active Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg. RIC will be conducted twice daily for 7 consecutive days.
  Interventions: Procedure: Remote ischemic conditioning
- Sham RIC (Placebo Comparator): Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg. RIC will be conducted twice daily for 7 consecutive days.
  Interventions: Procedure: Sham remote ischemic conditioning

INTERVENTIONS:
Procedure: Remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 200 mm Hg.
  Arms: RIC
Procedure: Sham remote ischemic conditioning — Remote ischemic conditioning (RIC) is induced by 4 cycles of 5 min of healthy upper limb ischemia followed by 5 min reperfusion. Limb ischemia was induced by inflation of a blood pressure cuff to 60 mm Hg.
  Arms: Sham RIC

SUMMARY:
The purpose of this study is to determine the impact of remote ischemic conditioning on cerebral hemodynamics in patients with ischemic stroke.

DETAILED DESCRIPTION:
Current studies have shown that remote ischemic conditioning can activate neuronal signals and humoral factors, increase cerebral perfusion and promote neurological recovery in patients with ischemic stroke.The purpose of this study was to investigate the effect of remote ischemic conditioning on cerebral hemodynamics in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, <80 years, both sex;
2. Patients with a clinically definite diagnosis of acute ischemic stroke who are able to commence RIC treatment within 72 hours of stroke onset;
3. Baseline National Institute of Health Stroke Scale (NIHSS) score<25;
4. Pre-onset modified Rankin Scale (mRS) score ≤ 1;
5. Glasgow Coma Scale score ≥8;
6. Signed and dated informed consent is obtained.

Exclusion Criteria:

1. Patients who have undergone thrombolytic therapy or endovascular therapy;
2. Inability to cooperate sufficiently to complete the cerebral autoregulation examination (e.g., due to a condition such as agitation, drowsiness, arrhythmia, insufficient bilateral temporal bone windows, etc.) during the recording;
3. Presence of other intracranial lesions, such as cerebrovascular malformations, cerebral venous thrombosis, tumors, and other brain lesions;
4. severe hepatic and renal dysfunction or failure;
5. Patients with hematological disease, abnormal coagulation function, bleeding tendency, and platelet <100×10^9/L;
6. Individuals who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper extremities, venous thrombosis in the acute or subacute stage of upper extremities, arterial occlusive disease, subclavian artery stenosis ≥ 50%, or subclavian steal syndrome;
7. pregnant or lactating women;
8. Previous RIC treatment or similar treatment;
9. Patients with a life expectancy of less than 3 months or patients who are unable to complete the study for other reasons;
10. unwillingness to be followed up or poor treatment adherence;
11. Individuals who are participating in other clinical studies, have participated in other clinical studies within 3 months prior to enrollment, or have participated in this research;
12. Other conditions that the investigator considers inappropriate for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral autoregulation at 7 days | 0 - 7 days
  Difference in Cerebral autoregulation at 7 days after RIC/sham-RIC between two groups. Phase difference (PD) in degree can therefore serve as a useful tool in the evaluation of cerebral autoregulation. Continuous cerebral blood flow velocities (CBFV) in cm/s of bilateral middle cerebral artery will be assessed noninvasively using transcranial Doppler. Spontaneous arterial blood pressure (ABP) in mmHg will be simultaneously recorded using a servo-controlled plethysmograph on the left or right middle finger with an appropriate finger cuff size. Data on CBFV and ABP were processed using MATLAB using scripts developed by the research team. PD was then derived from transfer function analysis to assess the dynamic association between CBFV and ABP.

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China